CLINICAL TRIAL: NCT03460132
Title: The Biological Effects of Commercial Orthodontic Miniscrews on the Oral Investing Tissue
Brief Title: Biological Effects of Commercial Orthodontic Miniscrews
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed S.M. Ammar, Assistant lecturer, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Al-Azhar 201
Record Dates: First submitted 2018-02-25; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Cytotoxicity
Keywords: orthodontic miniscrews; biological effect; cytotoxicity; metal release

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extraction cases (Experimental): patients receive Tomas orthodontic miniscrew implant as a mean of anchorage augmentation
  Interventions: Device: Tomas® Anchorage System - DENTAURUM

INTERVENTIONS:
Device: Tomas® Anchorage System - DENTAURUM — self drilling, bone inserted, screw like device used for anchorage preparation during orthodontic treatment.

SUMMARY:
The use of miniscrew implants as an anchorage device in orthodontics has gained a widespread acceptance in recent years. There prevailed use has been attributed to its ease in insertion and removal at a relatively low cost with no need to wait for a long time between miniscrew insertion and force application. In this regard; clinical studies have suggested that miniscrew implants may provide stable anchorage during the orthodontic treatment without requiring patient cooperation. These studies proved many successful applications in orthodontics involving; retraction of anterior teeth, correction of open bites, distalization, mesialization, and intrusion of teeth

DETAILED DESCRIPTION:
The use of miniscrew implants as an anchorage device in orthodontics has gained a widespread acceptance in recent years. There prevailed use has been attributed to its ease in insertion and removal at a relatively low cost with no need to wait for a long time between miniscrew insertion and force application. In this regard; clinical studies have suggested that miniscrew implants may provide stable anchorage during the orthodontic treatment without requiring patient cooperation. These studies proved many successful applications in orthodontics involving; retraction of anterior teeth, correction of open bites, distalization, mesialization, and intrusion of teeth.

In dentistry, various materials are used in implant systems. The implant material must be nontoxic, biocompatible, mechanically sufficient, and having high tension and corrosion resistance. Commercially pure titanium (cp Ti) is the most used material in prosthetic implants because of its; high biocompatibility, high corrosion resistance in body fluids, not allergic, high specific strength, and low elastic modulus when compared with other metallic biomaterials.

On the other hand, orthodontic miniscrew implants are smaller than conventional prosthetic implants and should resist high orthodontic loads. These factors contribute to the possible fracture of cp Ti miniscrew implants during placement, use, and removal. To avoid such fracture, Ti alloy implants, composed with aluminum (6Al) and vanadium (4V), (Ti-6Al-4V), for adding strength and fatigue resistance than cp Ti, are required. Unfortunately, this alloy has a low corrosion resistance and can result in corrosion of the orthodontic miniscrew implants in body fluids.

Any metal or alloy implanted in the human body is a potential source of toxicity. In an oral envelope, miniscrew implants are exposed to a number of potentially destructive physical and chemical agents. Evaluation the potential of conventional dental implants to release metallic ions into the body have been done. However, little attention has been given to metallic ion released from orthodontic miniscrew implant systems and the potential toxicity of these released metal on oral tissues. The concern about this has been limited to orthodontic brackets and wires.

One of the studies concerned with the biocompatibility of different metals used in vivo of different fixed orthodontic appliances and evaluating the presence of metal ions in oral mucosa cells, their potential cytotoxicity, and genotoxic effects. This study concluded that nickel and cobalt metals released from fixed orthodontic appliances could induce DNA damage in oral mucosa cells.

Literature review in this topic listed an expanding area of articles dealing with orthodontic miniscrews. The in vivo studies of cytotoxic effect of metal ions released from orthodontic miniscrew implants in body fluids are limited compared to in vitro studies.

In view of the above review of literature, it will be of great value in clinical orthodontics to investigate the biological effect of commercial orthodontic miniscrew implants on the oral investing tissue.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be included in this study if they have the following:

  1. All cases indicated for bilateral extraction of maxillary first premolar and retraction of canine into the extraction space.
  2. Age range from 14 to 18 years.
  3. Full set of permanent teeth (the third molars are not considered).
  4. No previous orthodontic or orthognathic surgery treatment.
  5. Good oral and general health.
  6. All teeth should be caries-free.
  7. All teeth should be free from any metallic restorations.

Exclusion Criteria:

* The patients will be excluded from the study if they have the following:

  1. History of serious medical problems or taking systemic medication which could affect orthodontic treatment.
  2. History of serious dental problems (endodontic treatment, apicectomy, or any other dental problems) which could affect orthodontic treatment.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
cytotoxicity of orthodontic miniscrew implant | 4 months after initiation of the orthodontic canine retraction
  Time dependent change in the percentage (%) of dead cells in series of swab samples harvested from area around orthodontic miniscrew implant.

SECONDARY OUTCOMES:
Metal release of orthodontic miniscrew implant | 4 months after initiation of the orthodontic canine retraction
  Time dependent change in the amount (micro-grams, µg) of titanium, aluminum and vanadium traces in series of saliva samples using inductively coupled plasma optical emission spectrometry.
surface changes of orthodontic miniscrew implants | 4 months after initiation of the orthodontic canine retraction
  surface analysis of orthodontic miniscrew implant (mass percentage) by X-ray fluorescence

IPD SHARING:
Plan to Share IPD: Undecided